CLINICAL TRIAL: NCT02565875
Title: Does Standardizing Language in Laparoscopic Surgery Improve Efficiency? A Randomized Controlled Trial
Brief Title: Standardizing Language in Laparoscopic Surgery
Acronym: SLL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Glenn Posner, Dr. Glenn D. Posner, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 20150727-01H
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Procedure Time; Communication
Keywords: Efficiency, Organizational; Simulation; Communication; Laparoscopy; Medical Education
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLL Presentation (Experimental): Intervention: Standardized Language of Laparoscopy (SLL) Presentation and simulated laparoscopic task performed on a low-fidelity pelvis simulator
  Will witness a presentation on the use of a SLL for communication between the primary and assistant surgeons during laparoscopy as previously determined by a national survey of Canadian experts and a modified delphi technique.
  Interventions: Behavioral: SLL Presentation; Other: Simulated laparoscopic task
- Control Presentation (Placebo Comparator): Intervention: Surgical Anatomy (SA) Presentation and simulated laparoscopic task performed on a low-fidelity pelvis simulator
  Will witness a presentation of similar duration as the intervention group on laparoscopy but not related to communication (laparoscopic anatomy). The simulated laparoscopic task will be identical to the SLL group.
  Interventions: Behavioral: Control Presentation; Other: Simulated laparoscopic task

INTERVENTIONS:
Behavioral: SLL Presentation — Educational presentation on the use of a standardized lexicon for communication between surgeon and assistant during laparoscopy
  Arms: SLL Presentation
Behavioral: Control Presentation — Educational presentation on relevant anatomy related to laparoscopy performed by a gynecologic surgeon.
  Arms: Control Presentation
Other: Simulated laparoscopic task — Using a low-fidelity pelvis simulator and laparoscopic instruments, pairs of each arm will be asked to perform a laparoscopic task (maneuver a ball into a nylon surgical bag). Use of SLL will be tabulated and task will be timed.

SUMMARY:
Obstetrics and Gynecology residents, fellows and attending physicians will be randomized to view one of two educational presentations of equal duration. The "intervention" presentation will demonstrate the use of a standardized language for effective communication of laparoscopy commands. Both groups will be asked to perform a simulated laparoscopic task. Participants will be timed and use of the standardized language will be tracked and tabulated. The primary outcome of interest is whether the use of standard commands during a simulated laparoscopic task is associated with sooner completion of the task. This may translate into improved efficiency in the operating room.

DETAILED DESCRIPTION:
Background

Continuous communication between the primary surgeon and assistant(s) during laparoscopic surgery is essential. The primary surgeon is rarely in direct control of the laparoscope and visual field. The use of a standard vernacular during surgery to provide clear instructions across all surgical centers is currently not employed. As the theoretical benefits of this are clear, a national survey produced a lexicon of commands1. Despite making intuitive sense, there is presently no evidence to demonstrate a benefit from using this standardized language during laparoscopic surgery. We aim to show that in doing so, there will be a significant improvement in speed and efficiency when performing a complex laparoscopic task.

Objective

To explore whether standardization of communication between the primary surgeon and the assistant in a simulated laparoscopic environment decreases the time needed to perform a complex task.

Materials and Methods

All subjects will provide demographic data, which will be collected through a brief questionnaire. This questionnaire will collect information regarding level of training or years of practice, as well as handedness. Personal identifying information (PII) will not be collected.

Subjects will be block randomized into control and intervention groups by random number generation. Block randomization will preserve equivalent distribution of level of training or years in practice into each group. Secondarily, handedness will be evenly distributed among groups, but not superseding level of training or years in practice.

The intervention group will receive a presentation on the standardized laparoscopic lexicon (SLL) (Mehdizadeh et al). The presentation will focus on sections 1-3 (surgical roles, camera commands and instrument commands).

The control group will receive no pre-task presentation.

Members within each group will be assigned a laparoscopic trainer by random allocation (blinded selection of card denoting station assignment). Through this, each trainer will have 2 subjects of the same group randomly assigned to it. These subjects will be referred to as the "primary surgeon" and "assistant". Assignment of initial roles will be done randomly. A member in each pair will be assigned the role denoted on a card he/she chooses blindly.

Pairs will be provided the task of placing a ball into a bag and closing the opening through tensioning the drawstring. This task must be performed using only laparoscopic graspers and will be timed by invigilators.

The ball will be approximately the same diameter as the bag opening and large enough to require camera adjustments. This task is not a commonly practiced laparoscopic skill such as suturing or knot tying (therefore should be less influenced by level of training) and should require communication between "primary surgeon" and "assistant" to accomplish in a timely fashion. The task is complex and should require sufficient time to detect a difference between groups.

Data collection within each group will include each pair's time to completion of the task and level of training/years in practice of "primary surgeon" and "assistant". Invigilators will track the usage of SLL during the task in both groups.

After a break, the roles will be reversed and the task repeated. The same data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Obstetrics and Gynecology Residents OR fellows OR attending physicians

Exclusion Criteria:

* Physical disability preventing the candidate from performing laparoscopic surgery

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Procedure Time | Recorded once per simulated laparoscopic task upon completion (one visit)
  The simulated laparoscopic task will be timed from initiation to completion

SECONDARY OUTCOMES:
Communication | Recorded during per simulated laparoscopic task (one visit)
  Tabulated instances of the use of SLL during simulated laparoscopic task from initiation to completion

OTHER OUTCOMES:
Post-Intervention Survey | After completion of simulated laparoscopic task (one visit)
  Survey requesting qualitative data on experience and the effect of presentations on anxiety during simulated task

CONTACTS AND LOCATIONS:
Overall Officials: Glenn D Posner, MDCM, FRCSC, Principal Investigator — Medical Director of the University of Ottawa Skills and Simulation Centre
Locations (1):
- University of Ottawa Skills and Simulation Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared, but will be available upon request as it will not contain any identifying data on the participant as determined through our institution's IRB.

REFERENCES:
- [Result] Mehdizadeh, Mehra, et al. Standardizing Language in Laparoscopy: A Modified Delphi Approach. (Poster) AIME Day, The University of Ottawa, Canada